CLINICAL TRIAL: NCT02750371
Title: Effect of Irradiation of the Cavernous Sinus and the Sellar Region on Autobiographical Memory
Acronym: ISOMAB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CHUBX 2015/03
Record Dates: First submitted 2016-04-20; First posted 2016-04-25 (Estimated); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Cavernous Sinus Meningioma; Pituitary Adenoma
Keywords: Cavernous sinus meningioma; Pituitary adenoma; Hippocampus; Irradiation; Autobiographical memory
MeSH Terms: conditions — Pituitary Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients with brain tumors treated by radiotherapy (Experimental): Patients with:
  - meningioma of the cavernous sinus for which radiotherapy is planned
  Or
  - a pituitary adenoma for which radiotherapy is planned
  Interventions: Other: Evaluation of autobiographical memory

INTERVENTIONS:
Other: Evaluation of autobiographical memory — Patients will answer several questionnaires one and two years after irradiation treatment end.

SUMMARY:
Several studies showed that radiotherapy as brain tumors treatment may affect cognition. It was observed that durable memory impairments could arise at irradiated patients if radiotherapy is applied on medial temporal lobes.

However, results concerned studies of anterograde memory and none, this day, estimates the impact of radiotherapy on autobiographical memory which also involves hippocampus.

The aim of this study is to evaluate effects of cavernous sinus or sellar region irradiation on autobiographical memory.

Thirty 35 to 65 years old patients, with cavernous sinus meningioma or pituitary adenoma for who radiotherapy is indicated will be recruited.

DETAILED DESCRIPTION:
Several studies showed that radiotherapy as brain tumors treatment may affect cognition. It was observed that durable memory impairments could arise at irradiated patients if radiotherapy is applied on medial temporal lobes. However, results concerned studies of anterograde memory and none, this day, estimates the impact of radiotherapy on autobiographical memory which also involves hippocampus, as specified in Nadel and Moscovitch model, the Multiple Trace Theory.

Autobiographical memory impairment issue is fundamental for identity construction. Prevent those impairments is important to quality of life improvement after such treatments.

The aim of this study is to evaluate effects of cavernous sinus or sellar region irradiation on autobiographical memory.

A pilot study was conducted with 10 patients affected by left cavernous sinus meningioma divided in two groups: the first one with untreated patients and the second one with patients who received cavernous sinus irradiation between 2 and 5 years before pilot study. This study indicated autobiographical memory deterioration in two groups and a worsening in treated group. Study limits did not allow us to draw conclusions. That is why, sample size will be extended and patients with cavernous sinus meningioma or pituitary adenoma will be recruited because of proximity between cavernous sinus, pituitary gland and hippocampus. Investigators wish to recruit 30 patients with cavernous sinus and meningioma.

Investigators hope for confirm our results from pilot study.

ELIGIBILITY:
Inclusion Criteria:

* Age between 35 and 65.
* Patient with:

  * meningioma of the cavernous sinus for which radiotherapy is planned
  * or a pituitary adenoma for which radiotherapy is planned
* French Mother tongue
* Person affiliated to national insurance
* Person who give its verbal agreement to participate

Exclusion Criteria:

* Presence of a serious psychiatric disorder (major depression, psychotic disorders, etc.) and central nervous system disease (epilepsy, multiple sclerosis, etc.).
* Treatment with chemotherapy
* General intellectual abilities deficient (IQ <80)
* Extension front of their meningioma
* Deficient Language Skills.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2016-07-27 (Actual); Primary Completion 2022-03 (Actual); Study Completion 2022-03 (Actual)

PRIMARY OUTCOMES:
Autobiographical memory test (TEMPau) score | Two years after irradiation treatment end

SECONDARY OUTCOMES:
Autobiographical memory test (TEMPau) score | One year after irradiation treatment end
Revised Self Consciousness Scale (RSCS) score | One and two years after irradiation treatment end
Quality of life questionnaire (QLQC-30/BN20) score | One and two years after irradiation treatment end
California Verbal Learning Test (CVLT) score | One and two years after irradiation treatment end

CONTACTS AND LOCATIONS:
Overall Officials: Olivier BRANCHARD, Study Chair — University Hospital, Bordeaux
Locations (1):
- University Hospital Bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No
Patient could request investigator an access to IPD according to French regulation (act No. 78-17 of 6 January 1978 on data processing, data files and individual liberties, amended by act No. 2004-801 of 6 August 2004).

REFERENCES:
- [Background] Nadel L, Moscovitch M. Memory consolidation, retrograde amnesia and the hippocampal complex. Curr Opin Neurobiol. 1997 Apr;7(2):217-27. doi: 10.1016/s0959-4388(97)80010-4. PMID 9142752
- [Background] Cabeza R, St Jacques P. Functional neuroimaging of autobiographical memory. Trends Cogn Sci. 2007 May;11(5):219-27. doi: 10.1016/j.tics.2007.02.005. Epub 2007 Mar 26. PMID 17382578
- [Background] Mizumatsu S, Monje ML, Morhardt DR, Rola R, Palmer TD, Fike JR. Extreme sensitivity of adult neurogenesis to low doses of X-irradiation. Cancer Res. 2003 Jul 15;63(14):4021-7. PMID 12874001